CLINICAL TRIAL: NCT02563262
Title: Human Neutral Body Posture in Weightlessness
Acronym: HYDRONAUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-122
Record Dates: First submitted 2015-07-22; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- body angles measurements during weightlessness (Other): body angles : ankle, knee, hip, shoulder, elbow, wrist, and neck.
  Interventions: Other: body angles measurements during weightlessness

INTERVENTIONS:
Other: body angles measurements during weightlessness

SUMMARY:
The scientific goal of this experiment is to evaluate the performances of our three-dimensional digital model by comparing its prediction computed from underwater data to posture observed during real weightlessness during parabolic flight.

DETAILED DESCRIPTION:
Investigations description Throughout the experiment test subject will be safely attached to a fixation mechanism at its center of gravity (hip). This mechanism comprises a climbing harness connected to two lateral vertical guides by two magnetic connection plates at the level of the hips. The test subject will lie down on the floor on a plate equipped with foam pads to create a comfortable lying surface. This mechanism allows free postural movement in microgravity phase and also supports the test subject´s lying position during 1,8g- phase. At any stage of the experiment the test subject will be able to exit the fixation alone, by using one hand only.

The harness can be moved vertically by a linear sliding system and springs in the vertical guides. Springs will remain compressed during the 1g/2g-phase and lift the subject with the reduction to microgravity.

At the beginning of the weightlessness phase of each parabola, the sliding system will push participant's body up to about 30cm above the floor. After he has reached the free floating position, he will be asked to perform a short effort (crouching or stretching) and then to relax and stay still.

Once free floating, three video cameras with wide angle lenses will record body movements from front, side and top view. By electronically synchronizing the cameras the produced images can be used for three-dimensional analysis. Additionally three-dimensional force sensors at the hip fixation will be used to evaluate the quality of microgravity provided during the parabolic flight.

Experimental protocol Before flight subjects will be familiarized with the setup and the protocol. For each flight day, 3 subjects will be studied. The procedure will be the same for the 3 subjects and on all 3 days.

The subject rests calm at the bottom until microgravity phase starts. As described above a spring forced linear sliding system will push his body mass up to about 300mm. After the test subject has reached its free floating position without any contact to the surrounding area (bottom), he will perform a short effort (crouching or stretching). From now on the subject should relax and is not allowed to move his muscles intentionally. At the end of microgravity phase, the sliding system will allow a soft landing on the foam pads.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude .There will be no additional test performed for subject selection.
* Who already participated in a underwater test in Munich

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Joint angles | baseline
  Angles of several joints (ankle, knee, hip, shoulder, elbow, wrist, and neck) measured with video cameras

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France